CLINICAL TRIAL: NCT01852695
Title: A Family Integrated Care Model For The Neonatal Intensive Care Unit: A Cluster Randomised Controlled Trial
Brief Title: Family Integrated Care in the NICU
Acronym: FICare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Foothills Medical Centre (Other); Sunnybrook Health Sciences Centre (Other); London Health Sciences Centre (Other); St. Boniface Hospital (Other); CHU de Quebec-Universite Laval (Other); IWK Health Centre (Other); Hamilton Health Sciences Corporation (Other); The Hospital for Sick Children (Other); Horizon Health Network (Other); Regina General Hospital (Other); Royal University Hospital Foundation (Other); Windsor Regional Hospital (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); The Moncton Hospital (Unknown); Health Sciences Centre, Winnipeg, Manitoba (Other); Kingston Health Sciences Centre (Other); Victoria General Hospital (Unknown); Janeway Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 122173
Record Dates: First submitted 2012-12-19; First posted 2013-05-14 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2015-10

CONDITIONS: Premature Birth
Keywords: Family integrated Care; Family centered care; NICU family centered care; NICU parent program
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Integrated Care Arm (Experimental): Parents are integrated into the care of their infants in the NICU. Parents consent to spending up to eight hours a day with their infant, attend special education sessions, participate in daily medical rounds, and do basic infant charting. This will enable parents to provide care for infants with nursing supervision in the areas of feeding, bathing, dressing and holding skin to skin.
  Interventions: Behavioral: Family Integrated Care
- Control Arm (No Intervention): Regular care by nurse will be provided to patients admitted to control sites.

INTERVENTIONS:
Behavioral: Family Integrated Care — Parents are integrated into the care of their infants in the NICU. Parents consent to spending up to eight hours a day with their infant, attend special education sessions, participate in daily medical rounds, and do basic infant charting. This will enable parents to provide care for infants with nursing supervision in the areas of feeding, bathing, dressing and holding skin to skin.
  Arms: Family Integrated Care Arm

SUMMARY:
In the highly technological environment of the modern neonatal intensive care unit (NICU), the infant is physically, psychologically and emotionally separated from its parents. Recognition that this impedes parent- infant interaction and is detrimental to the infant, led to the development of programs such as family centered care, kangaroo care and skin-to-skin care1-3. However, they are based on the common premise that only NICU professionals with special skills can provide care for the infant. Parents are relegated to a supportive role, and some have described themselves as voyeurs who are "allowed" to visit and hold their infants4. Many feel anxious and unprepared to care for their infants after discharge5.

In 1979, a shortage of NICU nurses in Estonia prompted Levin1,6 to implement a "humane" care model in which parents provided nursing care for the infant (except for administration of IV fluid and medication), while nurses provided teaching and guidance to parents. This resulted in 30% improvement in weight gain1,30% reduction in infections, 20% reduction in NICU length of stay, 50% reduction in nurse utilization and overall improved satisfaction among parents and staff [personal communication, Levin,A.]. Building on the Estonian experience, we have developed a new Family Integrated Care (FIC) model that is adapted for the NICU environment in North America. In a pilot study at Mount Sinai Hospital, Toronto 46 infants and their families were enrolled in the study. Preliminary results and feedback from parents and healthcare providers (HCP) show that the FIC model is both feasible and safe, and may lead to improved outcomes including improved weight gain(paper submitted for publication). This study is a cluster randomized controlled trial in 16 tertiary level NICUs, to evaluate the efficacy of the FIC model in Canada.

ELIGIBILITY:
Inclusion Criteria:

* < 33 weeks gestational age at birth;
* On no respiratory support or low level respiratory support (i.e., oxygen by cannula or mask, or continuous positive airway pressure (CPAP);
* A primary caregiver parent who is willing and able to commit to spending at least 8 hours per day with her/his infant between the hours of 0700 and 2000;
* Parental consent.

Exclusion Criteria:

* Palliative care;
* Major life threatening congenital anomaly;
* Critical illness (unlikely to survive);
* On high level of respiratory support (mechanical ventilator, high frequency oscillatory or jet ventilation, extra-corporeal membrane oxygenation)
* Parental request for early transfer to another hospital;
* Parental inability to participate (e.g., health, social or language issues that might inhibit their ability to communicate with the healthcare team).

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2013-03; Primary Completion 2015-10 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Weight Gain | Day 0-21
  Change in weight from enrollment to day 21 following commencement of the intervention

SECONDARY OUTCOMES:
Weight gain velocity | Day 0-21
  Weight gain velocity at 21 days post-intervention commencement;
Breastfeeding rate | up to 16 weeks
  Participants will be followed until first discharge home from hospital, an expected average 13 weeks
Clinical outcomes (mortality and Nosocomial infection (NI), Necrotizing Enterocolitis (NEC), Bronchopulmonary Dysplasia(BPD), Retinopathy of prematurity(ROP) & Intraventricular haemorrhage(IVH) | up to 16 weeks
  Patients will be followed for the duration of their hospital stay for an expected average of 13 weeks. Mortality and five major morbidities: (a) Nosocomial infection will be defined using the Center for Disease Control criteria; (b) Necrotizing enterocolitis is defined using Bell's criteria;(c) Bronchopulmonary dysplasia is defined according to Shennan et al; (d) Intraventricular hemorrhage will be classified using the Canadian Pediatric Society classification, from cranial ultrasound performed during the first 28 days of life; (e) Retinopathy of prematurity will be staged according to the International Classification of Retinopathy of Prematurity.
Safety | 1000 patient days
  Number of critical incident reports/1000 patient days
Parental stress and anxiety | Day 0 and when the infant reaches 35 weeks corrected gestational age
  We will administer questionnaires to parents in the first week following admission and when their infant reaches 35 weeks corrected gestational age, in both the intervention and control sites
Resource Use | Day 0 -week 16
  Data on health care utilisation will be collected during the patients entire hospital stay until the first discharge home, averaging 13 weeks including length of stay, duration of oxygen therapy. Per diem costs will be used to estimate potential cost savings derived from any reduced length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Shoo K Lee, FRCPC PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (15):
- Canada (15):
  - Foothills Medical Centre, Calgary, Alberta
  - Health Sciences Centre, Winnipeg, Winnipeg, Manitoba
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - IWK Health Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Centre hospitalier universitaire de Québec, Laval, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mclean MA, Scoten OC, Yu W, Ye XY, Petrie J, Church PT, Soraisham AS, Mirea LS, Weinberg J, Synnes AR, O'Brien K, Grunau RE. Lower Maternal Chronic Physiological Stress and Better Child Behavior at 18 Months: Follow-Up of a Cluster Randomized Trial of Neonatal Intensive Care Unit Family Integrated Care. J Pediatr. 2022 Apr;243:107-115.e4. doi: 10.1016/j.jpeds.2021.12.055. Epub 2021 Dec 29. PMID 34971651
- [Derived] Synnes AR, Petrie J, Grunau RE, Church P, Kelly E, Moddemann D, Ye X, Lee SK, O'Brien K; Canadian Neonatal Network Investigators; Canadian Neonatal Follow-Up Network Investigators. Family integrated care: very preterm neurodevelopmental outcomes at 18 months. Arch Dis Child Fetal Neonatal Ed. 2022 Jan;107(1):76-81. doi: 10.1136/archdischild-2020-321055. Epub 2021 Jun 18. PMID 34145042
- [Derived] O'Brien K, Robson K, Bracht M, Cruz M, Lui K, Alvaro R, da Silva O, Monterrosa L, Narvey M, Ng E, Soraisham A, Ye XY, Mirea L, Tarnow-Mordi W, Lee SK; FICare Study Group and FICare Parent Advisory Board. Effectiveness of Family Integrated Care in neonatal intensive care units on infant and parent outcomes: a multicentre, multinational, cluster-randomised controlled trial. Lancet Child Adolesc Health. 2018 Apr;2(4):245-254. doi: 10.1016/S2352-4642(18)30039-7. Epub 2018 Feb 8. PMID 30169298
- [Derived] O'Brien K, Bracht M, Robson K, Ye XY, Mirea L, Cruz M, Ng E, Monterrosa L, Soraisham A, Alvaro R, Narvey M, Da Silva O, Lui K, Tarnow-Mordi W, Lee SK. Evaluation of the Family Integrated Care model of neonatal intensive care: a cluster randomized controlled trial in Canada and Australia. BMC Pediatr. 2015 Dec 15;15:210. doi: 10.1186/s12887-015-0527-0. PMID 26671340